CLINICAL TRIAL: NCT03082794
Title: Investigating the Effects of Negative Calorie Diet Compared With Low-Calorie Diet on Weigh Loss and Lipid Profile in Sedentary Overweight/Obese Middle-Aged and Older Men
Brief Title: Dietary Effects on Weight Loss and Lipid Profile in Sedentary Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P.L.Shupik National Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, MD, PhD, Asst. Prof. of sports medicine (sports injury and corrective movement), University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: no Grant 4
Record Dates: First submitted 2017-03-04; First posted 2017-03-17 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Men; Life Style; Lipid Metabolism Disorders; Obesity; Overweight
Keywords: Dietary Formulations; Lifestyle; Obesity; Overweight; weight loss
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Lipid Metabolism Disorders; Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group I (Experimental): Study group I (53 participants) received the NCD (details of diet: 15% protein, 75% carbohydrates, 10% fat). Both groups had 15% caloric restriction from their maintenance energy requirements.
  Interventions: Dietary Supplement: NCD
- Study group II (Experimental): Study group II (51 participants) received the LCD or healthy weight maintenance diet (details of diet: 15% protein, 55% carbohydrates, 30% fat).Both groups had 15% caloric restriction from their maintenance energy requirements.
  Interventions: Dietary Supplement: LCD

INTERVENTIONS:
Dietary Supplement: NCD — Negative Calorie Diet
  Other Names: group I
  Arms: Study group I
Dietary Supplement: LCD — Low Calorie Diet
  Other Names: group II
  Arms: Study group II

SUMMARY:
Negative-calorie diet is among the popular dieting guides for weight loss; however, there is still little knowledge about this method. The present study aimed to determine the effects of negative-calorie diet on weight loss and lipid profile, and to compare its efficiency with low-calorie diet in men.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Weight-stable (± 2 kg, for more than one year)
* No history of regular exercise (in at least three months before the study).

Exclusion Criteria:

* History of medical disorders (CVD and other such as diabetes, depression, eating disorders, chronic medications, kidney disease, cancer, food allergies or intolerances to items used in meals, abnormality in thyroid or Electrocardiograph
* History of anti-obesity medication or weight loss drugs or dietary supplementations for weight control.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants were non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.
Enrollment: 104 (Actual)
Dates: Start 2011-02-20 (Actual); Primary Completion 2012-09-20 (Actual); Study Completion 2012-12-27 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline
  assessed in kg
Total cholesterol (Total-C) | Baseline
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | Baseline
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | Baseline
  assessed in mg/dl
Triglycerides (TG) | Baseline
  assessed in mg/dl

SECONDARY OUTCOMES:
Weight | 3-month
  assessed in kg
Total cholesterol (Total-C) | 3-month
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | 3-month
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | 3-month
  assessed in mg/dl